CLINICAL TRIAL: NCT00536276
Title: Vitamin D Deficiency in Acutely Injured Pediatric Burn Patients: Incidence, Etiology, Metabolic Sequelae and Prevention
Brief Title: Evaluation of Vitamin D Status in Children With Acute Burns
Acronym: VitaminD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Director, Nutrition Services, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-9-26-1
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Burns; Bone Demineralization
Keywords: vitamin D
MeSH Terms: conditions — Burns; Bone Demineralization, Pathologic | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Vitamin D2 — Daily enteral dose of 100IU/kg
  Other Names: ergocalciferol
Dietary Supplement: Vitamin D3 — Daily enteral dose of 100IU/kg
  Other Names: cholecalciferol

SUMMARY:
To see which vitamin D supplement (D2 vs D3) is most beneficial in burned children.

DETAILED DESCRIPTION:
The purpose of this study is to follow up our descriptive observations with a prospective randomized double blinded study to verify our clinical perception that hypovitaminosis D is prevalent postburn and to evaluate whether therapeutic supplementation will enhance specific primary outcome measures during burn convalescence.

ELIGIBILITY:
Inclusion Criteria:

* Child is > 6 months of age but < 19 years old
* Burn injury > 30% total body surface area
* Admitted to SHC within 4 days of injury
* Attending physician decision that patient is likely to survive
* Parents or legal guardian give informed consent along with assent of the child as applicable

Exclusion Criteria:

* Attending physician decision that patient is not likely to survive
* Prior history of anticonvulsant or glucocorticoid use, gastric/bowel resection, parathyroid disease, liver disease, chronic renal failure or prior pharmacologic vitamin D use (>1000 IU/D)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2003-03; Primary Completion 2009-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Examine the effect of D2 vs D3 supplementation on serum 25-OH and 1,25 OH vitamin D levels | During acute phase postburn

SECONDARY OUTCOMES:
Identify the most efficacious vitamin D analogue in terms of preventing deterioration of bone markers | During acute phase postburn

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gottschlich, PhD, RD, CNSD, Principal Investigator — Shriners Hospital for Children
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Gottschlich MM, Mayes T, Khoury J, Warden GD. Hypovitaminosis D in acutely injured pediatric burn patients. J Am Diet Assoc. 2004 Jun;104(6):931-41, quiz 1031. doi: 10.1016/j.jada.2004.03.020. PMID 15175591
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842